CLINICAL TRIAL: NCT02309671
Title: A Randomised, Controlled, Assessor-blind, Parallel Groups, Multicentre Trial Assessing the Dose-response Relationship of FE 999049 in Controlled Ovarian Stimulation in Japanese Women Undergoing an Assisted Reproductive Technology Programme
Brief Title: A Dose-response Trial Using FE 999049 in Japanese Women Undergoing in Vitro Fertilisation (IVF) / Intracytoplasmic Sperm Injection (ICSI) Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000124
Record Dates: First submitted 2014-11-28; First posted 2014-12-05 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2016-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — FE 999049; follitropin beta

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (4):
- FE 999049 6 µg (Experimental)
  Interventions: Drug: FE 999049
- FE 999049 9 µg (Experimental)
  Interventions: Drug: FE 999049
- FE 999049 12 µg (Experimental)
  Interventions: Drug: FE 999049
- FOLLISTIM 150 IU (Active Comparator): follitropin beta
  Interventions: Drug: follitropin beta

INTERVENTIONS:
Drug: FE 999049
  Arms: FE 999049 12 µg; FE 999049 6 µg; FE 999049 9 µg
Drug: follitropin beta
  Other Names: FOLLISTIM
  Arms: FOLLISTIM 150 IU

SUMMARY:
This trial investigates the effects of several doses of FE 999049 in Japanese women undergoing IVF/ICSI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with tubal infertility, unexplained infertility, infertility related to endometriosis stage I/II or with partners diagnosed with male factor infertility
* Women eligible for IVF and/or ICSI treatment
* Women aged 20-39 years
* Women with body mass index (BMI) of 17.5-32.0 kg/m2

Exclusion Criteria:

* Women with polycystic ovary syndrome (PCOS) associated with anovulation, endometriosis stage III/IV
* Women with history of recurrent miscarriage
* Women with contraindications to controlled ovarian stimulation with gonadotropins
* Women with three or more controlled ovarian stimulation cycles

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | End of stimulation (max 16 days after investigational medicinal product (IMP) start)

SECONDARY OUTCOMES:
Number of follicles during stimulation | Up to 16 days
Size of follicles during stimulation | Up to 16 days
Endocrine profile measured by circulating levels of hormones | Up to 16 days
Total IMP dose administered measured from first until last dose (end of stimulation) | Up to 16 days
Embryo quality measured by fertilised oocytes and number and quality of embryos and blastocysts during culturing | 5 days (from oocyte retrieval to embryo transfer)
Successful pregnancy rate | 5-6 weeks after transfer
Frequency of adverse events | From signing informed consent form until end of trial visit = 8-9 weeks
Intensity of adverse events | From signing informed consent form until end of trial visit = 8-9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Investigational site (there may be other sites in this country), Tokyo, Japan

REFERENCES:
- [Result] Ishihara O, Klein BM, Arce JC; Japanese Follitropin Delta Phase 2 Trial Group. Randomized, assessor-blind, antimullerian hormone-stratified, dose-response trial in Japanese in vitro fertilization/intracytoplasmic sperm injection patients undergoing controlled ovarian stimulation with follitropin delta. Fertil Steril. 2021 Jun;115(6):1478-1486. doi: 10.1016/j.fertnstert.2020.10.059. Epub 2020 Dec 4. PMID 33272623